CLINICAL TRIAL: NCT01717196
Title: Diagnostic Accuracy of FNA (Fine Needle Aspiration) on Solid Pancreatic Lesions: is Aspiration- Related?
Brief Title: Diagnostic Accuracy of FNA: is Aspiration- Related?
Acronym: expect fna
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EX0001
Record Dates: First submitted 2012-10-22; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: PANCREATIC CANCER
Keywords: sample adequacy; diagnostic accuracy; complications
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DIFFERENT VOLUME ASPIRATION BIOPSY (Experimental): The needle system was in all cases the 22 gauge EUS-FNA (Expect needle). After the puncture the stylet was removed, and we performed three punctures with a 22 G needle with both volume aspiration 10 and 20 cc and without syringe for each lesion. The sequence of different volume aspiration Biopsy/ FNA (10cc, 20cc, no aspiration) was randomly assigned by sealed envelope system.
  Interventions: Other: different volume aspiration

INTERVENTIONS:
Other: different volume aspiration — comparison between diagnostic yield of FNA on solid pancreatic masses performed with different aspiration volume (10 and 20ml) and without aspiration.

SUMMARY:
BACKGROUND: EUS-FNA has a central role in the diagnostic algorithm of solid pancreatic masses. Different needle diameters and the use of stylet are not associated with differences in terms of diagnostic yield for malignancy. Preliminary studies showed that using suction (10ml) is associated with a higher sensitivity for cancer diagnosis. We aim to compare EUS-FNA in the same solid pancreatic mass performed with the 22 gauge needle with different aspiration volumes (10, 20, 0ml), looking for adequacy, diagnostic accuracy and complications.

METHODS: Prospective clinical study at four referral Centers: ISMETT Palermo; Bellaria-Maggiore, Bologna; Civico-A.R.N.A.S, Palermo; Humanitas-IRCCS, Rozzano. EUS was performed by five experienced echo-endoscopist. The needle system was in all cases the 22 gauge EUS-FNA(Expect). We performed three punctures with a 22 G needle with both volume aspiration 10 and 20 cc and without syringe for each lesion. The sequence (10cc, 20cc, no aspiration) was randomly assigned by sealed envelope system. For each pass tissue samples were smeared into slides for ROSE(Rapid-On-Site-Evaluation); after smearing sample into the slides, the material was fixed in formalin for cyto-histological evaluation. The cyto-pathologist was always blinded as to which aspiration was used for which specimen. After EUS-FNA the patients were monitored for at least six hour to detect immediately post-procedural complication and were followed up during the 30 days post-procedure in order to detect late complications.

DETAILED DESCRIPTION:
Background

EUS-FNA has a central role in the diagnostic algorithm of solid pancreatic masses [ASGE Practice Committee] with high sensitivity and specificity (75-92% - 82-100%), [1-2-3] and low complication rate (1-2%) [4-5-6]. In the clinical setting of solid pancreatic mass a histological diagnosis appears highly relevant both for differential diagnosis (adenocarcinoma, lymphoma or neuroendocrine tumour) and for optimal therapeutic decision. For the cythopathologic diagnosis of pancreatic cancer, sensitivity increased with the operator's experience and reached 80% after 20 to 30 EUS-FNA. Furthermore it well demonstrated that on-site cytopathology interpretation during the procedure increase the diagnostic yield of EUS-FNA [7-8]. ROSE (Rapid On -Site Evaluation) may be useful to guide the number of FNA passes, learn which parts of the lesion may be targeted for increased diagnostic yield, and correct technical errors (e. g. bloody or paucicellular material) [9, 10]. The diagnostic yield of EUS-guided biopsies depends on size, location and characteristics of target tissues as well as on technical and procedural factors (type of needle, biopsy technique and material processing) [11-20].

Expertise and training of endosonographer and interaction with the cytopathologist have also an important role [7-14-15]. Up to now three different sizes of needle are available for collecting cytological material: 25 - 22 and 19 gauge with an aspiration volume syringe of 10ml. Most of the studies on EUS-FNA have been conducted using 22G needles. Data on thinner (25G) or larger (19G) needles are limited. A number of recent studies, including two RCTs, compared results obtained with needles of various diameters. All these studies were performed in the setting of pancreatic masses [18-20]. Although thinner needles provide less cellular material than do larger needles, the specimens from the former are less contaminated by blood, and thus easier to interpret. In addition, thinner needles may be easier to use because of greater flexibility, particularly for locations requiring important scope bending [18, 19]. An RCT in 131 patients found no significant differences between 22G and 25G needles in terms of diagnostic yield for malignancy [17]. Finally another RCT compared EUS-FNA without ROSE using 19G or 22G needles in 117 patients [18] showed a similar diagnostic accuracy for both needles.

If the diameter of the needle used does not appear to affect the diagnostic accuracy of FNA on solid pancreatic lesions, preliminary studies show that using suction during EUS FNA of solid masses is associated with a significantly higher sensitivity for cancer diagnosis (86% vs. 67%; P=0.05) [20]. A pilot trial suggested that applying continuous high pressure suction (using a balloon inflation device) allowed retrieval of tissue samples for histopathological examination in most cases [21].

A new needle Expect by Boston Scientific are available with an aspiration syringe with variable volume of 5-10-15-20cc. No studies were performed comparing the diagnostic yield of FNA on solid pancreatic masses performed with different aspiration volume (10 and 20ml) and without aspiration.

Aims

The aims of our prospective study are to compare EUS-FNA in the same solid pancreatic mass performed with the 22 gauge needle with aspiration volume syringe of 10ml, 20ml and without aspiration, looking for: sample adequacy, diagnostic accuracy, complications.

Methods

Patients This was a prospective clinical study at four referral center for EUS: ISMETT/UPMC (Mediterranean Institute for Transplantation and Advanced Specialized Therapies/University of Pittsburgh Medical Center in Italy), Palermo; AUSL Bologna, Bellaria-Maggiore Hospital; Civico-A.R.N.A.S. Hospital, Palermo; Humanitas IRCCS, Rozzano, Milano. We planned to collect at least 100 cases in 3 months. The study protocol conforms to the ethical guidelines of the 1975 Declaration of Helsinki (6th revision, 2008) as reflected in a priori approval by the institution's human research committees.

The inclusion criteria for the study were: diagnosed or suspected solid pancreatic lesions according to imaging (CT-scan or/and MRI); no contraindications for FNA (see exclusion criteria). The exclusion criteria were: age < 18 years; cystic pancreatic lesions; history of previous gastrectomy; patients hemodynamically unstable or with severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 60.000 cells/cubic millimetre [cmm3]); patients unable to suspend anticoagulant therapy; pregnancy; inability to give informed consent; refusal to participate to the study.

Data on comorbidity and chronic treatment were recorded as well as data on possible complications related to the procedure. Patients undergoing anticoagulant or antiaggregant therapy for noncritical problems discontinued the treatment at least 5 days before the endoscopic procedure or until INR normalization, starting low dose heparin. Written informed consent was obtained from all patients for the procedures performed. All procedures were performed under conscious sedation with meperidine ± midazolam or deep sedation with propofol according to each center guideline and patient clinical condition.

Procedure Endoscopic ultrasonography was performed using a linear echo-endoscope by five experienced echo-endoscopist with a current case volume of at list 500 per year (200 FNA). The standard technique for FNA was adopted: the needle is advanced under real-time EUS guidance into the target lesion by using a quick, strong thrust of the handle. The stylet is completely withdrawn and a syringe attached to the end of the needle device. Once inside the lesion, after applying negative pressure suction by opening the lock device of the syringe, the needle is moved back and forth 15 times under EUS guidance. The suction syringe is then released, the needle withdrawn into the catheter, and the whole system removed from the echoendoscope.

The needle system was in all cases the 22 gauge EUS-FNA (Expect needle). After the puncture the stylet was removed, and we performed three punctures with a 22 G needle with both volume aspiration 10 and 20 cc and without syringe for each lesion. The sequence (10cc, 20cc, no aspiration) was randomly assigned by sealed envelope system.

Technical success was defined as puncturing the target tissue properly without technical difficulties (inability of the needle to exit from the channel of the scope) or mechanical rupture and obtaining some visible tissue specimens or fragments with each puncture.

Tissue samples was immediately smeared into slides after each puncture, fixed and all the prepared slides will be viewed by experienced pathologists for ROSE (Rapid On Site Evaluation). For each pass, after smearing sample into the slides, the material was fixed in formalin for cyto histological evaluation. The cytopathologist was always blinded as to which aspiration was used for which specimen.

The cases will be stratified into 4 diagnostic categories applied for ROSE and for histological evaluation:

a) Positive for malignancy, b) Suspicious for malignancy, c) Negative for malignancy, d) Non diagnostic.

For each aspiration two fundamental parameters will be evaluated on slides and formalin fixed sample: sample adequacy intended as overall cellularity (including normal, neoplastic, non-epithelial cells) and diagnostic accuracy.

Post-procedural follow-up After EUS-FNA the patients were monitored for at least six hour to detect immediately post-procedural complication and were followed up with a scheduled protocol during the 30 days post-procedure in order to evaluate clinical status, blood chemistry, and to detect late complications. All patients were followed up for at least 1 month. All adverse events were evaluated and related or not to the procedure. All data were recorded electronically on excel database for the final analysis.

STATISTICAL ANALYSIS Data were analyzed using the SPSS 15 software package (SPSS Inc., Chicago, Illinois, USA). Continuous variables were summarized as means ± SD, or range, when appropriate. Categorical variables were summarized as frequency and percentage. For comparison of qualitative variables, a chi-squared test was calculated. For comparison of quantitative variables, Students t test was used. Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall accuracy for each arm was investigated. Differences were considered significant at a P value of <0.05 (two-sided).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed or suspected solid pancreatic lesions according to imaging (CT-scan or/and MRI);
* no contraindications for FNA (see exclusion criteria).

Exclusion Criteria:

* age < 18 years;
* cystic pancreatic lesions;
* history of previous gastrectomy;
* patients hemodynamically unstable or with severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 60.000 cells/cubic millimetre [cmm3]);
* patients unable to suspend anticoagulant therapy;
* pregnancy;
* inability to give informed consent;
* refusal to participate to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
sample adequacy | 20min
  Tissue samples was immediately smeared into slides after each puncture, fixed and all the prepared slides will be viewed by experienced pathologists for ROSE (Rapid On Site Evaluation). For each pass, after smearing sample into the slides, the material was fixed in formalin for cyto histological evaluation. The cytopathologist was always blinded as to which aspiration was used for which specimen.

SECONDARY OUTCOMES:
diagnostic accuracy | 5 days
  For each pass, after smearing sample into the slides, the material was fixed in formalin for cyto histological evaluation. The cytopathologist was always blinded as to which aspiration was used for which specimen.
  The cases will be stratified into 4 diagnostic categories applied for ROSE and for histological evaluation:
  a) Positive for malignancy, b) Suspicious for malignancy, c) Negative for malignancy, d) Non diagnostic.

OTHER OUTCOMES:
complications | up to 30 days after the procedure
  After EUS-FNA the patients were monitored for at least six hour to detect immediately post-procedural complication and were followed up with a scheduled protocol during the 30 days post-procedure in order to evaluate clinical status, blood chemistry, and to detect late complications. All patients were followed up for at least 1 month. All adverse events were evaluated and related or not to the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria tarantino, MD, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- ISMETT, Palermo, Italy